CLINICAL TRIAL: NCT03476304
Title: Comparison of Endocrowns Longevity and Post Retained Restorations: Randomized Clinical Trial
Brief Title: Endocrown Restorations Longevity Compared With Post Retained Restorations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Maximiliano Sergio Cenci, PhD, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PPGO023
Record Dates: First submitted 2018-03-14; First posted 2018-03-26 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Endodontically Treated Teeth
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Semi-direct composite endocrown restorations (Experimental)
  Interventions: Device: Endocrown restoration
- Post retained direct composite restoration (Active Comparator)
  Interventions: Device: Post retained composite restoration
- Post retained ceramic restoration (Active Comparator)
  Interventions: Device: Post retained ceramic restoration

INTERVENTIONS:
Device: Endocrown restoration — The endodontically treated tooth will be impressed, and an endocrown restoration will be manufactured with resin composite in a cast and cemented with self adhesive cement
  Arms: Semi-direct composite endocrown restorations
Device: Post retained composite restoration — The endodontically treated tooth will receive a fiber post cemented with self adhesive cement and after this, the tooth will be impressed and a semi direct composite restoration will be cemented with self adhesive cement.
  Arms: Post retained direct composite restoration
Device: Post retained ceramic restoration — The endodontically treated tooth will receive a fiber post cemented with self adhesive cement and after this, the tooth will be impressed and a ceramic restoration will be cemented with self adhesive cement.
  Arms: Post retained ceramic restoration

SUMMARY:
Caries disease is still the leading cause of severe tooth decay. Since this can lead to tooth loss, it is important that appropriate treatment is advised to help prevent damage and maintain tooth health. Faced with major coronary destruction, several times it becomes necessary to perform the endodontic treatment, aiming to maintain the element in the buccal cavity for longer. It is known that an excellent restorative treatment with poor endodontic treatment and the inverse has a direct impact on the (in) success of the treatment. In this context, the proper cleaning of the root canals is highlighted, aiming the removal of bacteria and toxins. Acceptable restorations are those that provide adequate reestablishment of anatomy, function, proximal contacts, and occlusal stability. Traditionally, indirect restorations would be indicated in cases of extensive coronary destruction, because it was believed that they would present greater resistance and longevity when compared to direct restorations. However, contemporary dentistry admits that, thanks to adhesive and conservative principles, this difference between direct and indirect procedures in terms of longevity is not significant. The classic restorative procedure in cases of endodontically treated teeth with great loss of coronary structure involves the use of intraradicular retainers, followed by the creation of core and restoration through total crowns. Removal of healthy tissue for the use of posts can weaken the remaining dental structure and increase the risk of root perforations. In this sense, endocrown restorations show superiority when compared to those made with intraradicular retainers. Although the indications are favorable for the use of endocrown restorations, the clinical evidence available on the subject is still scarce. In this double-blind randomized clinical trial, patients who need and meet the inclusion criteria will will be allocated to one of the three restorative groups available, being endocrown restoration in semi-direct composite resin, direct restoration in composite resin retained on the post and ceramic crown retained in the post. Patients will be monitored annually after completion of restorative treatment outcome. In addition to treatment longevity, other secondary outcomes will be evaluated, such as patient satisfaction, impact on quality of life and cost-effectiveness of the proposed treatments.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more;
* healthy volunteers;
* molars or premolars with endodontic treatment and large coronal destruction;
* at least 20 teeth;

Exclusion Criteria:

* abutment of removable partial denture ;
* tooth with mobility higher than 1;
* more than 1/2 bone loss height;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2018-04-02 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Survival | 2 years
  Tooth will be annually followed until failure, but with a minimal follow-up of two years. They will be evaluated with FDI criteria for evaluation of direct and indirect restorations

SECONDARY OUTCOMES:
Satisfaction and quality of life improvement | 2 years
  Questionnaire will be applied
Cost-effectiveness | 2 years
  The calculation of cost-effectiveness after treatment delivery will be performed

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Pelotas, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No